CLINICAL TRIAL: NCT02310126
Title: Handling Comparison Between Two Contact Lens Types
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: CR-5570
Record Dates: First submitted 2014-12-03; First posted 2014-12-05 (Estimated); Results first posted 2016-03-31 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2017-06

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- etafilcon A(sphere)/etafilcon A(multi-focal) (Active Comparator): Subjects were randomized to one of two lens wear sequences. subjects randomized to this sequence received etafilcon A (sphere) contact lens first and then the etafilcon A (multi-focal) contact lens second.
  Interventions: Device: etafilcon A (multi-focal); Device: etafilcon A (sphere)
- etafilcon A(multi-focal)/etafilcon A(sphere) (Active Comparator): Subjects were randomized to one of two lens wear sequences. subjects randomized to this sequence received etafilcon A (multi-focal) contact lens first and then the etafilcon A (sphere) contact lens second.
  Interventions: Device: etafilcon A (multi-focal); Device: etafilcon A (sphere)

INTERVENTIONS:
Device: etafilcon A (multi-focal) — Each subject will wear the soft contact lenses for 15 minutes then remove the lenses.
  Other Names: Investigational Multifocal Contact
Device: etafilcon A (sphere) — Each subject will wear the soft contact lenses for 15 minutes then remove the lenses.
  Other Names: 1-DAY ACUVUE® MOIST®

SUMMARY:
Subjects will evaluate each study lens in a random order. The lenses will be worn in both eyes for a short period.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must read, understand and sign the Statement of Informed Consent and receive a fully executed copy of the form.
2. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
3. The subject must be between 40 and 70 years of age.
4. The subject's vertex corrected spherical equivalent distance refraction must be in the range of +0.25 to +4.00 or plano to -6.00 in each eye.
5. The subject's refractive cylinder must be less than or equal to -0.75 D in each eye.
6. The subject's ADD power must be in the range of +0.75 D to +2.50 D in each eye.
7. The subject best corrected visual acuity of 20/20 -3 or better in each eye.
8. Subject must own a wearable pair of spectacles.
9. The subject must be an adaptable soft contact lens wearer in both eyes (i.e. worn lenses a minimum of 2 days per week for at least 8 hours per day, for 1 month or more of duration)
10. The subject must already be wearing a presbyopic contact lens correction (e.g. reading spectacles over contact lenses, multifocal or monovision contact lenses, etc.) or if not responded positively to at least one symptom on the "Presbyopic Symptoms Questionnaire".

Exclusion Criteria:

1. Currently pregnant or lactating (subjects who become pregnant during the study will be discontinued).
2. Any ocular or systemic allergies or diseases that may interfere with contact lens wear.
3. Any systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear.
4. Any ocular abnormality that may interfere with contact lens wear.
5. Use of any ocular medication, with the exception of rewetting drops.
6. Any previous intraocular surgery (e.g. radial keratotomy, photorefractive keratectomy (PRK), laser-assisted in situ keratomileusis (LASIK), etc.)
7. Any grade 3 or greater slit lamp finding (e.g. edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) which may contraindicate contact lens wear.
8. Any ocular infection or inflammation.
9. History of herpetic keratitis.
10. Any corneal distortion or irregular cornea.
11. History of binocular vision abnormality or strabismus.
12. Any infectious disease (e.g. hepatitis, tuberculosis) or contagious immunosuppressive disease (e.g. HIV).
13. Current history of diabetes.
14. Participation in any contact lens or lens care product clinical trial within 30 days prior to study enrollment.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2014-12-01 (Actual); Study Completion 2014-12-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Baymeadows Vision Center, Jacksonville, Florida
  - Eye Elements Eyecare, Jacksonville, Florida
  - Vistakon Research Clinic, Jacksonville, Florida
  - Golden Family Eyecare, Sarasota, Florida
  - Eye Associates of Winter Park, Winter Park, Florida
  - Central Ohio Eyecare, Columbus, Ohio
  - Optometry Group LLC, Memphis, Tennessee
  - Nashville Vision Associates, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study enrolled a total of 195 subjects. Of those enrolled, 4 subjects did not meet the eligibility criteria, and 191 subjects were dispensed study lenses. Of those dispensed, subjects 189 completed the study and 2 subjects were discontinued. Subjects were stratified as either Hyperops or Myopes based on their sphere power.
Groups:
- Etafilcon A(Multi-focal)/Etafilcon A(Sphere): Subjects were randomized to one of two possible lens wear sequences. Subjects first received the etafilcon A (sphere) contact lens and then received the etafilcon A (multi-focal) contact lens.
- Etafilcon A(Sphere)/Etafilcon A(Multi-focal): Subjects were randomized to one of two possible lens wear sequences. Subjects first received the etafilcon A (sphere) contact lens and then received the etafilcon A(multi-focal) contact lens.
Period: Period 1 (15 Minutes)
Arm/Group | Etafilcon A(Multi-focal)/Etafilcon A(Sphere) | Etafilcon A(Sphere)/Etafilcon A(Multi-focal)
Started | 94 | 97
Hyperopes | 38 | 33
Myopes | 56 | 64
Completed | 94 | 95
Not Completed | 0 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Violation | 0 | 1
Period: Period 2 (15 Minutes)
Arm/Group | Etafilcon A(Multi-focal)/Etafilcon A(Sphere) | Etafilcon A(Sphere)/Etafilcon A(Multi-focal)
Started | 94 | 95
Hyperopes | 38 | 32
Myopes | 56 | 63
Completed | 94 | 95
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The analysis population consists of subjects that were dispensed at least one study lens.
Groups:
- Etafilcon A(Multi-focal)/ Etafilcon A(Sphere): Subjects were randomized to one of two possible lens wear sequences. Subjects first received the etafilcon A(multi-focal) contact lens and then received the etafilcon A(sphere) contact lens.
- Etafilcon A(Sphere) / Etafilcon A(Multi-focal): Subjects were randomized to one of two possible lens wear sequences. Subjects first received the etafilcon A(sphere) contact lens and then received the etafilcon A(multi-focal) contact lens.
- Total: Total of all reporting groups
Arm/Group | Etafilcon A(Multi-focal)/ Etafilcon A(Sphere) | Etafilcon A(Sphere) / Etafilcon A(Multi-focal) | Total
Number analyzed (Participants) | 94 | 97 | 191
Age, Continuous [Mean (Standard Deviation); unit: years]
  Hyperopes, N=38, N=33, N=71 | 55.2 (7.49) | 57.3 (6.45) | 56.2 (7.06)
  Myopes, N=56, N=64, N=120 | 50.8 (7.03) | 51.1 (7.24) | 51.0 (7.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 83 | 153
  Male | 24 | 14 | 38
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian Or Alaska Native | 1 | 0 | 1
  Asian | 0 | 1 | 1
  Black of African American | 4 | 8 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  White | 89 | 87 | 176
Region of Enrollment [Number; unit: participants]
  United States | 94 | 97 | 191

OUTCOME MEASURES:

1. Primary Outcome: Overall Lens Handling Using the Contact Lens User Experience(CLUE) TM Questionnaire.
Description: CLUE Overall Lens Handling is assessed using the Contact Lens User Experience (CLUE)TM questionnaire. CLUE is a validated patient-reported outcomes questionnaire to assess patient experience attributes of soft, disposable contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Scores follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response. 97% of the scores fall within 0 and 120 (mean +/-3XSD).
Time Frame: 15 minutes post Contact Lens Insertion
Population: The analysis population consist of subjects that completed all study visits without a major protocol deviation. The analysis was conducted for each lens and strata.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Etafilcon A(Multi-focal): Subjects that received the etafilcon A (multi-focal) contact lens during either the first or second period of the study.
- Etafilcon A (Sphere): Subjects that received the etafilcon A (sphere) contact lens during either the first or second period of the study.
Arm/Group | Etafilcon A(Multi-focal) | Etafilcon A (Sphere)
Number analyzed (Participants) | 184 | 184
units on a scale
  Hyperopes, N=69, N=69 | 53.44 (25.482) | 55.81 (26.432)
  Myopes, N=115, N=115 | 61.70 (24.594) | 60.23 (23.369)

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study (approximately 1 month)
Groups:
- Etafilcon A (Multi-focal): Subjects that received the etafilcon A (multi-focal) contact lens during either the first or second period of the study.
Arm/Group | Etafilcon A (Multi-focal) | Etafilcon A (Sphere)
Serious Adverse Events (participants affected / at risk) | 0/191 | 0/191
Other Adverse Events (participants affected / at risk) | 0/191 | 0/191

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days